CLINICAL TRIAL: NCT05812755
Title: The Effects of Soluble Guanylyl Cyclase Stimulation on Perioperative Vascular Reactivity and Organ Injury in Cardiac Surgery
Brief Title: SGC Stimulation, Perioperative Vascular Reactivity, and Organ Injury in Cardiac Surgery
Acronym: SOLSTICE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marcos G. Lopez, Associate Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 222089; R01HL164909 (NIH)
Record Dates: First submitted 2023-03-28; First posted 2023-04-14 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Endothelial Dysfunction; Vascular Diseases; Kidney Injury; Brain Disease; Vascular Inflammation
MeSH Terms: conditions — Vascular Diseases; Brain Diseases | interventions — vericiguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vericiguat (Active Comparator): 10 mg vericiguat administered orally once daily for three days (through day of surgery)
  Interventions: Drug: Vericiguat
- Placebo (Placebo Comparator): placebo administered orally once daily for three days (through day of surgery)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat — Vericiguat 10 mg administered orally starting 2 days prior to heart surgery through the day of surgery
  Arms: Vericiguat
Drug: Placebo — Matched placebo administered orally starting 2 days prior to heart surgery through the day of surgery
  Arms: Placebo

SUMMARY:
The goal of this mechanistic clinical trial is to learn about the effects of medications called soluble guanylyl cyclase stimulators on vascular function and markers of kidney and brain injury in patients having heart surgery. The main questions it aims to answer are:

1. Does soluble guanylyl cyclase stimulation improve blood vessel function compared to placebo?
2. Does soluble guanylyl cyclase stimulation decrease markers of kidney injury and brain injury compared to placebo?

Participants will be randomized to a soluble guanylyl cyclase stimulator called vericiguat or placebo, and researchers will compare vascular function and markers of brain and kidney injury to see if vericiguat improves vascular function and reduces markers of injury.

This will provide important information to determine the underlying reasons that patients have some kidney and brain function problems after having heart surgery.

DETAILED DESCRIPTION:
Patients undergoing elective cardiac surgery will be randomized to the soluble guanylyl cyclase stimulator vericiguat versus placebo before surgery through the day of surgery and vascular function will be quantified using ultrasound and direct assessment of arterial relaxation ex-vivo. Markers of brain and kidney injury will be measured in plasma and urine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Elective open-heart surgery, defined as surgery on the heart or aorta that requires sternotomy or thoracotomy

Exclusion Criteria:

1. Intolerance to vericiguat
2. Use of other soluble guanylyl cyclase stimulators or current use of phosphodiesterase-5 inhibitors
3. Pregnancy or breast feeding. Pregnancy will be excluded in women of child-bearing potential by a urine or serum beta hcg test
4. Renal replacement therapy within 30 days prior to screening
5. Estimated glomerular filtration rate <15 ml/min per 1.73 m2 per Chronic Kidney Disease Epidemiology collaboration (CKD-EPI) equation at time of screening
6. Systolic blood pressure less than 120 mmHg at the time of screening
7. Prior kidney transplantation
8. History of significant liver dysfunction (defined as Child-Pugh class C)
9. Surgery scheduled to be performed with circulatory arrest
10. Surgery scheduled to correct a major congenital heart defect
11. Extracorporeal membrane oxygenation (ECMO) prior to surgery
12. Active systemic infection or surgery for infectious endocarditis
13. Ventricular assist device or intraaortic balloon pump support prior to surgery
14. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | Day of surgery
  Percent change in brachial artery diameter from baseline to maximum post-forearm ischemia adjusted for shear-rate (Aim 1 primary outcome).
Ex vivo vascular relaxation | Day of surgery
  Ex vivo arterial relaxation (percent) in participants with available vascular tissue (Aim 1 primary outcome)
Ubiquitin C-terminal hydrolase L1 (UCHL1) plasma concentration | Enrollment through postoperative day 2
  UCHL1 will be measured in plasma to quantify effects of vericiguat vs. placebo on neuronal injury (Aim 2 primary neuronal outcome)
Neutrophil gelatinase associated lipocalin (NGAL) urine concentration | Enrollment through postoperative day 2
  NGAL will be measured in urine to quantify effects of vericiguat vs. placebo on markers of renal injury (Aim 2 primary renal outcome)

SECONDARY OUTCOMES:
Phosphorylated vasodilator stimulated phosphoprotein (phospho-VASP) | Enrollment through postoperative day 2
  Soluble guanylyl cyclase stimulation will be further quantified as arterial phospho-VASP/VASP ratio(Aim 1 secondary outcome)
Endothelial barrier breakdown - claudin-5 | Enrollment through postoperative day 2
  Endothelial barrier breakdown will be quantified as plasma concentration of claudin-5 (Aim 1 secondary outcome)
Endothelium mediated inflammation and coagulation - plasminogen activator inhibitor-1 (PAI-1) | Enrollment through postoperative day 2
  Endothelium mediated inflammation and coagulation will be quantified as plasma concentration of PAI-1 (Aim 1 secondary outcome)
Endothelial Activation - intercellular adhesion molecule 1 (ICAM1) | Enrollment through postoperative day 2
  Endothelial activation will be quantified as plasma concentrations of ICAM1 (Aim 1 secondary outcome)

OTHER OUTCOMES:
Exploratory clinical outcome: serum creatinine | Postoperative day 0 up to 1 year postoperatively (e.g., approximately 1 year after the day of surgery)
  Serum creatinine
Exploratory clinical outcome: Kidney Disease Improving Global Outcomes (KDIGO) Acute Kidney Injury (AKI) | Postoperative day 0 up to 1 year postoperatively (e.g., approximately 1 year after the day of surgery)
  Incidence of KDIGO creatinine criteria AKI
Exploratory clinical outcome: delirium | Postoperative day 0 to 10 days postoperatively
  Incidence (percent of participants) with a positive delirium exam measured using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).
Exploratory clinical outcome: delirium severity | Postoperative day 0 to 10 days postoperatively
  Severity of delirium measured using the CAM-ICU-7 score for at least 3 days postoperatively up to 10 days postoperatively for participants who remain in ICU. This is a 7 point scale score with higher scores indicating higher severity of delirium
Exploratory clinical outcome: Infection | Postoperative day 0 to 10 days postoperatively
  Infection defined as initiation of antibiotics postoperatively not part of perioperative antibiotic prophylaxis.
Exploratory clinical outcome: Respiratory failure | Postoperative day 0 to hospital discharge (e.g., up to approximately 30 days following surgery)
  Respiratory failure defined as the need for mechanical ventilation
Exploratory clinical outcome: Thrombocytopenia | Postoperative day 0 to hospital discharge(e.g., up to approximately 30 days following surgery)
  Thrombocytopenia defined at platelet count less than 50,000
Exploratory clinical outcome: Arrythmia | Postoperative day 0 to hospital discharge (e.g., up to approximately 30 days following surgery)
  Arrhythmia defined the onset of new atrial or ventricular dysrhythmia
Exploratory clinical outcome: Intensive care unit (ICU) length of stay | Postoperative day 0 to until discharge from the ICU (e.g. up to approximately 10 days following surgery)
  ICU length of stay in days
Exploratory clinical outcome: Hospital length of stay | Postoperative day 0 to hospital discharge (e.g., up to approximately 30 days following surgery)
  Hospital length of stay in days
Exploratory clinical outcome: Death | Postoperative day 0 to one year postoperatively
  Mortality measured up to one year
Exploratory cognitive status outcome: Telephone interview for cognitive status | 6 months postoperatively
  Six-month follow-up (Telephone Interview for Cognitive Status) obtained by phone interview. Maximum score is 41 and lower score indicates worse cognitive function.
Exploratory functional status outcome: Katz Activities of Daily Living (ADL) assessment | 6 months postoperatively
  Activities of daily living will be assessed with the Katz ADL assessment via phone interview. This survey assesses independence in 6 activities, and will be summarized as the average number of independent activities.
Exploratory functional status outcome: Pfeffer functional activities questionnaire | 6 months postoperatively
  Activities of daily living will be assessed with the Pfeffer functional activities questionnaire via phone interview. Maximum score is 30. A score of greater than 9 indicates impaired function and possible cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Lopez, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No